CLINICAL TRIAL: NCT01089010
Title: A Phase II, Double-Blind, Randomized, Placebo-Controlled, Three-Way Crossover, Pharmacokinetic and Pharmacodynamic Study of CK-2017357 in Patients With Amyotrophic Lateral Sclerosis (ALS)
Brief Title: A Study of CK-2017357 in Patients With Amyotrophic Lateral Sclerosis (ALS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cytokinetics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CY 4021
Record Dates: First submitted 2010-03-16; First posted 2010-03-18 (Estimated); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — CK-2017357

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Treatment Sequence 1 (Experimental): Treatment sequence 1 consisted of three dosing periods in which patients received single oral doses of placebo, 250 mg, and 500 mg of CK-2017357, in that order, with approximately one week between each dose. Each patient acted as their own control, as all doses were represented in each treatment sequence.
  Interventions: Drug: Placebo; Drug: 250 mg CK-2017357; Drug: 500 mg CK-2017357
- Treatment Sequence 2 (Experimental): Treatment sequence 2 consisted of three dosing periods in which patients received single oral doses of placebo, 500 mg, and 250 mg of CK-2017357, in that order, with approximately one week between each dose. Each patient acted as their own control, as all doses were represented in each treatment sequence.
  Interventions: Drug: Placebo; Drug: 250 mg CK-2017357; Drug: 500 mg CK-2017357
- Treatment Sequence 3 (Experimental): Treatment sequence 3 consisted of three dosing periods in which patients received single oral doses of 250 mg, placebo and 500 mg of CK-2017357, in that order, with approximately one week between each dose. Each patient acted as their own control, as all doses were represented in each treatment sequence.
  Interventions: Drug: Placebo; Drug: 250 mg CK-2017357; Drug: 500 mg CK-2017357
- Treatment Sequence 4 (Experimental): Treatment sequence 4 consisted of three dosing periods in which patients received single oral doses of 250 mg, 500 mg and placebo of CK-2017357, in that order, with approximately one week between each dose. Each patient acted as their own control, as all doses were represented in each treatment sequence.
  Interventions: Drug: Placebo; Drug: 250 mg CK-2017357; Drug: 500 mg CK-2017357
- Treatment Sequence 5 (Experimental): Treatment sequence 5 consisted of three dosing periods in which patients received single oral doses of 500 mg, placebo, and 250 mg of CK-2017357, in that order, with approximately one week between each dose. Each patient acted as their own control, as all doses were represented in each treatment sequence.
  Interventions: Drug: Placebo; Drug: 250 mg CK-2017357; Drug: 500 mg CK-2017357
- Treatment Sequence 6 (Experimental): Treatment sequence6 consisted of three dosing periods in which patients received single oral doses of 500 mg, 250 mg, and placebo of CK-2017357, in that order, with approximately one week between each dose. Each patient acted as their own control, as all doses were represented in each treatment sequence.
  Interventions: Drug: Placebo; Drug: 250 mg CK-2017357; Drug: 500 mg CK-2017357

INTERVENTIONS:
Drug: Placebo — Matching placebo in capsules administered as a single oral dose.
Drug: 250 mg CK-2017357 — 250 mg CK-2017357 in capsules administered as a single oral dose.
  Other Names: tirasemtiv
Drug: 500 mg CK-2017357 — 500 mg CK-2017357 in capsules administered as a single oral dose.
  Other Names: tirasemtiv

SUMMARY:
The primary objective of this study is to demonstrate a pharmacodynamic effect of CK 2017357 on measures of skeletal muscle function or fatigability in patients with ALS.

DETAILED DESCRIPTION:
This study is a Phase II, double-blind, randomized, placebo-controlled, three-way crossover study of CK-2017357 in patients with ALS. 36 to 72 patients will be randomized to one of six different treatment sequences. Each treatment sequence consists of three dosing periods; in each dosing period¸ patients receive a single oral dose of placebo, 250 mg of CK-2017357, or 500 mg of CK-2017357. All six treatment sequences will enroll approximately the same number of patients. A washout period of at least 6 days (to a maximum of 10 days) will be employed between the doses for each patient. This study is designed to assess the effect of CK-2017357 on maximal voluntary muscle strength, on the development of fatigue at maximal and sub-maximal voluntary muscle contraction, and on selected pulmonary function parameters. The plasma concentration of CK-2017357 will be measured at selected time points after each of two single doses of CK-2017357 in men and women. The plasma concentration versus time data obtained in this study may be used to develop a population PK model and estimate inter-subject variability of PK parameters in this target patient population, in particular between male and female study patients.

ELIGIBILITY:
Inclusion Criteria

For enrollment, patients were required to satisfy all of the following criteria at baseline:

1. Able to comprehend and willing to sign an Informed Consent Form (ICF)

1. A diagnosis of familial or sporadic ALS (defined as meeting the possible, laboratory-supported probable, probable, or definite criteria for a diagnosis of ALS according to the World Federation of Neurology El Escorial criteria) (Brooks, Miller et al. 2000)
2. Males or females 18 years of age or older
3. Body Mass Index (BMI) of 18.0 to 30.0 kg/m2, inclusive
4. Maximum voluntary grip strength in at least one hand between 10 and 40 pounds (females) or 10 and 60 pounds (males)
5. Able to swallow capsules with water
6. Upright Slow Vital Capacity (SVC) > 40% of predicted for age, height, and sex [See Appendix 16.6.1]
7. Able to perform pulmonary function tests
8. Pre-study clinical laboratory findings (including troponin I [TnI] and creatine phosphokinase [CPK]) within normal range, or, if outside of the normal range, deemed not clinically significant by the Investigator
9. For female patients only: The patient is post-menopausal (≥ 1 year) or sterilized, or if she is of childbearing potential, she is not breastfeeding, her pregnancy test is negative, she has no intention to become pregnant during the course of the study, and she is using contraceptive drugs or devices for the duration of the study and for 10 weeks after the end of the study.

For male patients only: Male patients agree for the duration of the study and 10 weeks after the end of the study to use a condom during sexual intercourse with female partners who are of reproductive potential and to have female partners use an additional effective means of contraception (e.g., diaphragm plus spermicide or oral contraceptives) or the male patient must agree to abstain from sexual intercourse for 10 weeks after the end of the study.

Exclusion Criteria

Patients satisfying any of the following criteria at baseline were excluded from enrollment:

1. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 3 times the upper limit of normal (ULN)
2. Life expectancy < 3 months
3. Participation in any trial in which receipt of investigational study drug occurred within 30 days prior to dosing
4. Any prior treatment with CK-2017357
5. In the opinion of the Investigator, the patient is not suitable to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2010-03; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
ALSFRS-R | 2 days
  An instrument for evaluating the functional status of patients with ALS. Minimum score is 0 and maximum score is 40. The higher the score the more function is retained.
Maximum grip strength | 2 days
  Measured using the DynEx Electronic Hand Dynamometer. Patients asked to squeeze the device with the maximum possible force to establish the maximum voluntary contraction.
Maximum grip strength fatigability | 2 days
  Handgrip fatigue is measured using the DynEx Electronic Hand Dynamometer. Patient is asked to squeeze the device until they can no longer stay above 60% of target or 120 seconds.
Shoulder extension fatigue | 2 days
  Patient is asked to hold one arm outstretched in front of them at a 90 degree angle. The time the arm falls below 90 degrees for > 2 seconds will be recorded, up to a total evaluation time of 2 minutes. This is then repeated with the other arm.
Slow Vital Capacity (SVC) | 2 days
  SVC is measured using the Puritan Bennett Renaissance II Spirometry System and accessories.
Maximum Voluntary Ventilation (MVV) | 2 days
  MVV is the volume of air that can be exhaled during 12 seconds of rapid deep breathing. The actual volume is extrapolated to one minute. the Puritan Bennett Renaissance II Spirometry System and accessories is used for this measurement.
Sniff Inspiratory Pressure (SNIP) | 2 days
  SNIP is measured at Functional Residual Capacity, the bottom of the tidal breathing cycle, through one plugged nostril while the other remains open using the Micro Medical MicroRPM Respiratory Pressure Meter
Maximum Voluntary Muscle Contraction (MVC) | 2 days
  MVC is measured using the MicroFET 2 HHD.
Repeated Sub-Maximum Grip Strength Fatigability | 2 days
  Sub-Maximum Grip Strength Fatigability is measured using the DynEx Electronic Hand. Dynamometer

SECONDARY OUTCOMES:
Characterize the relationship, if any, between the plasma concentration of CK-2017357 and ALSFRS-R. | 2 days
  ALSFRS-R assessments will be paired with PK concentrations obtained at or near the same time as the ALSFRS-R assessments and analyzed for concentration related effects.
Characterize the relationship, if any, between the plasma concentration of CK-2017357 and maximum grip strength | 2 days
  Maximum grip strength assessments will be paired with PK concentrations obtained at or near the same time as the maximum grip strength assessments and analyzed for concentration related effects.
Characterize the relationship, if any, between the plasma concentration of CK-2017357 and maximum grip strength fatigability | 2 days
  Maximum grip strength fatigability assessments will be paired with PK concentrations obtained at or near the same time as the maximum grip strength fatigability assessments and analyzed for concentration related effects.
Characterize the relationship, if any, between the plasma concentration of CK-2017357 and shoulder extension fatigue | 2 days
  Shoulder extension fatigue assessments will be paired with PK concentrations obtained at or near the same time as the shoulder extension fatigue assessments and analyzed for concentration related effects.
Characterize the relationship, if any, between the plasma concentration of CK-2017357 and slow vital capacity | 2 days
  Slow vital capacity assessments will be paired with PK concentrations obtained at or near the same time as the slow vital capacity assessments and analyzed for concentration related effects.
Characterize the relationship, if any, between the plasma concentration of CK-2017357 and maximum voluntary ventilation | 2 days
  Maximum voluntary ventilation assessments will be paired with PK concentrations obtained at or near the same time as the maximum voluntary ventilation assessments and analyzed for concentration related effects.
Characterize the relationship, if any, between the plasma concentration of CK-2017357 and sniff inspiratory pressure | 2 days
  Sniff inspiratory pressure assessments will be paired with PK concentrations obtained at or near the same time as the sniff inspiratory pressure assessments and analyzed for concentration related effects.
Characterize the relationship, if any, between the plasma concentration of CK-2017357 and maximum voluntary muscle contraction | 2 days
  Maximum voluntary muscle contraction assessments will be paired with PK concentrations obtained at or near the same time as the maximum voluntary muscle contraction assessments and analyzed for concentration related effects.
Characterize the relationship, if any, between the plasma concentration of CK-2017357 and repeated sub-maximum grip strength fatigability | 2 days
  Repeated sub-maximum grip strength fatigability assessments will be paired with PK concentrations obtained at or near the same time as the repeated sub-maximum grip strength fatigability assessments and analyzed for concentration related effects.
Number of patients with adverse events | 4 weeks
Effect of CK-2017357 on patient determined global functional assessment | 2 days
  Patients will be asked to assess whether they feel the same, better or worse as compared to how they felt pre-dose
Effect of CK-2017357 on investigator determined global functional assessment | 2 days
  Investigator will assess whether they the patient appears the same, better or worse as compared to the patient's status at pre-dose

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy M Shefner, MD, PhD, Study Chair — State University of New York - Upstate Medical University
Locations (15):
- United States (15):
  - Phoenix Neurological Associates, Ltd., Phoenix, Arizona
  - University Neurology Associates, Fresno, California
  - California Pacific Medical Center, San Francisco, California
  - Mayo Clinic Florida, Jacksonville, Florida
  - University of Kentucky, Lexington, Kentucky
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - SUNY Upstate Medical Center, Syracuse, New York
  - Duke University, Durham, North Carolina
  - Providence ALS Center, Portland, Oregon
  - Drexel University College of Medicine, Dept of Neurology, Philadelphia, Pennsylvania
  - Penn State, University Park, Pennsylvania
  - The University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Vermont, Burlington, Vermont

REFERENCES:
- [Result] Shefner J, Cedarbaum JM, Cudkowicz ME, Maragakis N, Lee J, Jones D, Watson ML, Mahoney K, Chen M, Saikali K, Mao J, Russell AJ, Hansen RL, Malik F, Wolff AA; Neals/Cytokinetics Study Team. Safety, tolerability and pharmacodynamics of a skeletal muscle activator in amyotrophic lateral sclerosis. Amyotroph Lateral Scler. 2012 Sep;13(5):430-8. doi: 10.3109/17482968.2012.684214. Epub 2012 May 16. PMID 22591195
- See also: Safety, tolerability and pharmacodynamics of a skeletal muscle activator in amyotrophic lateral sclerosis. — http://www.ncbi.nlm.nih.gov/pubmed/22591195